CLINICAL TRIAL: NCT04621058
Title: Efficacy of Treatment With Vitamin D in Patients Diagnosed With COVID-19 Who Presenting Vitamin D Deficiency and Pneumonia.
Brief Title: Efficacy of Vitamin D Treatment in Mortality Reduction Due to COVID-19.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioaraba Health Research Institute (Network)
Collaborators: Fundación Eduardo Anitua (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VITD
Record Dates: First submitted 2020-11-06; First posted 2020-11-09 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: SAR; SARS Pneumonia
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple-blind study, neither the patients, nor the researchers, nor those responsible for the statistical analysis will know the treatment that the patient is undergoing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D VITAMIN GROUP (Experimental): The administration of vitamin D will be carried out using the following treatment scheme:
  If vitamin D deficiency (< 30 ng/ml) treatment with 2 capsules of 0.266 mg If vitamin D deficiency (< 40 ng/ml): treatment with 1 capsule of 0.266 mg
  Blood levels of vitamin D will be determined on day 1, 4, 7 and 14. Based on the results from day 14, a new determination is recommended 4 weeks after starting treatment with the primary care physician who will decide whether to continue or interrupt the treatment. This phase will be carried out outside of the study.
  In addition, the product should only be administered, if blood calcium and phosphorus levels are within normal limits, as well as if the creatinuria/calciuria ratio is within normal ranges.
  Interventions: Drug: Vitamin D
- PLACEBO GROUP (Placebo Comparator): The procedure will be the same as in the experimental group but instead of the active component, patients will take placebo capsules exactly the same as above but without the active component.
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: Vitamin D — In case of Vitamin D levels <30 or 40ng/ml patients will take vitamin D supplements.
  Other Names: D VITAMIN GROUP
  Arms: D VITAMIN GROUP
Drug: PLACEBO — Placebo capsules exactly the same as the above, but without the active component.
  Other Names: PLACEO GROUP
  Arms: PLACEBO GROUP

SUMMARY:
HYPOTHESIS: The administration of vitamin D supplements to patients who have a positive diagnosis for SARS-Cov-2, acute pneumonia requiring hospital admission and vitamin D deficiency have a more favourable evolution than subjects not treated with vitamin D (placebo). This favourable evolution will translate into a reduction in mortality, fewer ICU admissions and fewer days of stay in hospital.

OBJECTIVES:

PRINCIPAL: To assess whether the group of patients receiving vitamin D supplements have a less severe evolution of their acute pneumonia, translated into lower mortality, than patients who do not receive that supplement.

SECONDARY: 1) To determine the number of intensive care admissions and the number of days of admission in both groups (control group and intervention group). 2) To estimate the prevalence of Vitamin D deficiency in the patients studied and the effectiveness of its supplementation. 3) To establish the degree of complexity of each study group and carry out a cost-effectiveness study.

METHODOLOGY: DESIGN: Clinical trial, randomized, placebo-controlled and double-blind, with two parallel groups The active treatment will be vitamin D (Hydroferol soft capsules of 0.266 mg). The placebo will consist of a tablet with the same external characteristics and with the same treatment scheme but which will not contain any vitamin D active ingredients.

DETAILED DESCRIPTION:
HYPOTHESIS: The administration of vitamin D supplements to patients who have a positive diagnosis for SARS-Cov-2, acute pneumonia requiring hospital admission and vitamin D deficiency have a more favourable evolution than subjects not treated with vitamin D (placebo). This favourable evolution will translate into a reduction in mortality, fewer ICU admissions and fewer days of stay in hospital.

OBJECTIVES:

PRINCIPAL: To assess whether the group of patients receiving vitamin D supplements have a less severe evolution of their acute pneumonia, translated into lower mortality, than patients who do not receive that supplement.

SECONDARY: 1) To determine the number of intensive care admissions and the number of days of admission in both groups (control group and intervention group). 2) To estimate the prevalence of Vitamin D deficiency in the patients studied and the effectiveness of its supplementation. 3) To establish the degree of complexity of each study group and carry out a cost-effectiveness study.

METHODOLOGY: DESIGN: Clinical trial, randomized, placebo-controlled and double-blind, with two parallel groups The active treatment will be vitamin D (Hydroferol soft capsules of 0.266 mg). The placebo will consist of a tablet with the same external characteristics and with the same treatment scheme but which will not contain any vitamin D active ingredients.

Inclusion criteria: Adult patients admitted to the Respiratory/Internal Medicine Unit of Santiago hospital of the OSI Araba HUA for acute pneumonia and suffering from a vitamin D deficit (< 30 ng/ml) and a RT-PCR, in nasopharyngeal exudate, positive for SARS-CoV-2.

Exclusion criteria: 1)Patients taking any type of vitamin D supplement. 2)Patients with hypoparathyroidism. 3) Patients in whom the administration of vitamin D is formally contraindicated. 4) Patients who cannot take vitamin D orally.

OUR SIZE: In order to answer to the main objective (mortality reduction 21% versus 50% intervention and control group respectively), we will need a total sample of 108 evaluable subjects-54 patients per group (J Crit Care. 2018;44:300-5).Statistical power 90%,95% statistical significance with possible loss of follow-up of 5% of patients.

A recruitment period of about 12 months is needed.

STATISTICAL ANALYSIS: In order to answer to the main and secondary objectives (mortality and ICU admission), the Chi-square test will be performed and in the event that any of the frequencies is less than 5, the exact Fisher test will be used.

Depending on the distribution of the quantitative variables, the Student t-test for independent samples or the non-parametric Mann-Whitney U-test will be used, respectively.

The analysis criterion will be "by intention to treat". In all cases. The statistical significance will be 95%.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the Respiratory or Internal medicine Units of Santiago hospital (HUA) due to pneumonia.
* Vitamin D deficiency (25(OH) defined by blood levels below 30 mg/ml.
* Possibility for observation during the treatment period.
* Signing of written consent (oral informed consent exceptionally).
* Positive PCR for diagnosis of sars-cov2 infection

Exclusion Criteria:

* Patients taking any type of vitamin D supplement.
* Patients with hypoparathyroidism.
* Pregnant or lactating women.
* Patients in whom the administration of vitamin D is formally contraindicated (see annex VI).
* Patients who at time of inclusion, cannot take vitamin D orally.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
MORTALITY | At 21 days.
  Mortality reduction

SECONDARY OUTCOMES:
Intensive care admissions | At 21 days
  Intensive care admissions reduction
Length of hospital stay | AT 21 DAYS
  Length of hospital stay reduction
Prevalence of vitamin D deficiency | At baseline
  To assess the prevalence of vitamin D deficiency at baseline
Incremental cost effectiveness ratio (ICER) | At 21 days
  To calculate the incremental cost per event (mortality) avoided

CONTACTS AND LOCATIONS:
Overall Officials: Joaquín Durán Cantolla, Principal Investigator — Bioaraba Health Research Institute
Locations (1):
- Joaquín Durán Cantolla, Vitoria-Gasteiz, Alava, Spain

IPD SHARING:
Plan to Share IPD: Undecided